CLINICAL TRIAL: NCT00055172
Title: The Determination of Genetic Basis Of Immunodeficiency
Brief Title: Genetic Basis of Immunodeficiency
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030105; 03-H-0105
Record Dates: First submitted 2003-02-20; First posted 2003-02-20 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12-04

CONDITIONS: Severe Combined Immunodeficiency
Keywords: Cytokines; Inherited Immunodeficiency; Natural History
MeSH Terms: conditions — Severe Combined Immunodeficiency

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-sibling relative: 18 years of age or older
- Patients (index cases): Patients (index cases), 6 months of age or older
- Siblings: Siblings, 6 months of age or older

SUMMARY:
This study will examine the role of hereditary factors in different forms of severe combined immunodeficiency (SCID).

Patients with immunodeficiencies may be eligible for this study. Candidates include:

* Patients with diminished numbers of T cells or NK cells or both, or
* Patients with normal T cell and NK cell numbers but diminished T cell, B cell, or NK cell function.

Relatives of patients will also be studied.

Participants will have blood samples collected for genetic analysis in studies related to SCID at the National Institutes of Health and other institutions.

DETAILED DESCRIPTION:
The goal of this project is to identify the genetic basis of new forms of inherited immunodeficiency. The particular focus relates to cytokines such as IL-2, IL-4, IL-7, IL-9, IL-15, and IL-21 that share the common cytokine receptor (Gamma) chain, (Gamma c), and to molecules that are important for signaling or gene regulation in response to these cytokines, although other causes of inherited immunodeficiency are also encompassed.

ELIGIBILITY:
* INCLUSION CRITERIA:

Index cases to be included are those with diminished numbers of T cells and/or NK cells and/or B cells or other immune cells or those who have normal numbers of T cell, B cells, NK cells and other immune cells but diminished function of one or more immune cells. Relatives of affected individuals may also be studied

* Patients (index cases): 6 months of age and older
* Siblings: 6 months of age and older
* Non-sibling relatives (biological parent, aunt, uncle or grandparent): 18 years or older

EXCLUSION CRITERIA:

* Patients with a known diagnosis
* Patients with a particular immunological phenotype that is not of interest to the research conducted under this study.
* Pregnancy or lactation
* Adults with current decisional impairment

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2004-04-05 (Actual)

PRIMARY OUTCOMES:
To identify forms of inherited immunodeficiency resulting from mutation of yc dependent cytokines, components of their receptors, or signaling molecules in their pathways | ongoing
  In an effort to determine the cause of the immunodeficiency, we will perform studies that may include but not be limited to evaluating the levels of expression of protein and/or mRNA, obtaining DNA sequence data, performing epigenetic studies, and evaluating biological function using cellular, biochemical, or other molecular studies.

CONTACTS AND LOCATIONS:
Overall Officials: Warren J Leonard, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Noguchi M, Yi H, Rosenblatt HM, Filipovich AH, Adelstein S, Modi WS, McBride OW, Leonard WJ. Interleukin-2 receptor gamma chain mutation results in X-linked severe combined immunodeficiency in humans. Cell. 1993 Apr 9;73(1):147-57. doi: 10.1016/0092-8674(93)90167-o. PMID 8462096
- [Background] Russell SM, Tayebi N, Nakajima H, Riedy MC, Roberts JL, Aman MJ, Migone TS, Noguchi M, Markert ML, Buckley RH, O'Shea JJ, Leonard WJ. Mutation of Jak3 in a patient with SCID: essential role of Jak3 in lymphoid development. Science. 1995 Nov 3;270(5237):797-800. doi: 10.1126/science.270.5237.797. PMID 7481768
- [Background] Puel A, Ziegler SF, Buckley RH, Leonard WJ. Defective IL7R expression in T(-)B(+)NK(+) severe combined immunodeficiency. Nat Genet. 1998 Dec;20(4):394-7. doi: 10.1038/3877. PMID 9843216
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2003-H-0105.html